CLINICAL TRIAL: NCT05796882
Title: Impact of the Whole Food Plant-Based Diet in HIV-Associated Reduction in Cardiovascular Risk
Brief Title: Whole Food Plant-Based Diet for HIV-Associated Reduction in Cardiovascular Risk (PLANT-HART)
Acronym: PLANT-HART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Chihuahua (Other)
Responsible Party: Principal Investigator, Carolina Martínez Loya, MD, Médico Pasante de Servicio Social, Universidad Autonoma de Chihuahua
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 023C-03/23; CI-023 (Other: Comité de Investigación del Hospital Central del Estado)
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Heart Diseases; Hiv
Keywords: HIV; Heart disease; Risk Factors; Plant-based; Cardiovascular
MeSH Terms: conditions — Heart Diseases; Acquired Immunodeficiency Syndrome | interventions — Diet, Vegan; Diet, Plant-Based; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Prospective study, randomized pilot clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention (type of diet) is not possible to mask either the participants or the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WFPBD Group (Experimental): The participants in this group follow a Whole Food Plant-Based Diet for 8 weeks
  Interventions: Behavioral: Whole Food Plant-Based Diet Ad Libitum
- Nutritional Standard Care Group (Active Comparator): The participants in this group receive a nutritional consultation every month with dietetic guidance and recommendations about a healthy lifestyle, duration 8 weeks
  Interventions: Behavioral: Nutritional Standard Care

INTERVENTIONS:
Behavioral: Whole Food Plant-Based Diet Ad Libitum — Participants will follow a Low Fat Whole Food Plant-Based Diet Ad Libitum for 8 weeks. It consists of increasing the daily consumption of fruits and vegetables, including sources of vegetable protein such as legumes (beans, lentils, chickpeas, peas, etc), soybeans and their derivatives (tofu, textured soybeans, soymilk), and whole grains. (oats, wheat, rice, quinoa, corn), nuts and seeds high in omega-3 fatty acids (chia, flaxseed, hemp), and minimize processed foods, and foods high in saturated fat. Avoiding animal-sourced foods.
  There will be no caloric restriction, however, visual support will be provided, in the form of a traffic light, to distinguish the frequency with which each type of food can be consumed
  Other Names: Vegan diet; Plant-based diet
  Arms: WFPBD Group
Behavioral: Nutritional Standard Care — Nutritional Consultation every month for 2 months. Recommendations on healthy eating and lifestyle will be given. Duration 8 weeks
  Other Names: Nutritional Counseling
  Arms: Nutritional Standard Care Group

SUMMARY:
The goal of this clinical trial is to evaluate the impact of using a whole food plant-based diet in the reduction of cardiovascular risk related to HIV in people who live with HIV infection.

The main questions it aims to answer are:

* Does a whole food plant-based diet, nonrestrictive in calories and low in fat, reduce the cardiovascular risk associated with HIV infection in people with HIV infection?
* Does the whole food plant-based diet permit achievement goals in specific metabolic markers of cardiovascular risk (such as Cholesterol, C Reactive Protein)? Participants will follow a non-calorie restricted, low fat, whole food plant-based diet for 8 weeks Researchers will compare standard nutritional care to see if there is a difference in the main outcomes

DETAILED DESCRIPTION:
The participants in the group within the intervention will follow a Whole Food Plant-Based Diet for 8 weeks, which consists of increasing the daily consumption of fruits and vegetables, including sources of vegetable protein such as legumes (beans, lentils, chickpeas, peas, etc. ), soybeans and their derivatives (tofu, textured soybeans, soymilk), and whole grains (oats, wheat, rice, quinoa, corn), nuts and seeds high in omega-3 fatty acids (chia, flaxseed, hemp ), minimize processed foods and foods high in saturated fat. There will be no caloric restriction, however, visual support will be provided, in the form of a traffic light, to distinguish the frequency with which each type of food can be consumed. A small recipe book will be provided with suggestions for breakfast, lunch, and dinner dishes. Patients will receive vitamin b12 supplements of 1000 micrograms twice a week.

There will be no caloric restriction, however, visual support will be provided, in the form of a traffic light, to distinguish the frequency with which each type of food can be consumed. A small recipe book will be provided with suggestions for breakfast, lunch, and dinner dishes. Patients will receive vitamin b12 supplements of 1000 micrograms twice a week.

The participants in the other group will attend a consultation with a nutritionist every month in which will receive recommendations about nutrition and lifestyle in order to reduce cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years but under 60 years
* Individuals with a BMI >25
* Individuals with some classic cardiovascular risk factor (dyslipidemia, smoking, type 2 diabetes mellitus, systemic arterial hypertension, obesity)
* Individuals under ART with adequate CD4+ cell count and viral load undetectable

Exclusion Criteria:

* Patients currently diagnosed with AIDS
* Patients who have suffered an AMI and/or stroke
* Patients who use drugs
* Patients who have had poor adherence to ART

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Risk | 8 weeks
  Estimate of the 10-year risk of myocardial infarction or death calculated by the Framingham score for coronary artery disease

SECONDARY OUTCOMES:
Systolic Blood Pressure | 8 weeks
  Maximum pressure exerted by the heart when it beats measured in mmHg
Percentage of body fat | 8 weeks
  Estimated percentage of fat mass using bioimpedance
LDL cholesterol | 8 weeks
  Type of lipoprotein measured in milligrams per deciliter
Percentage of body muscle mass | 8 weeks
  Estimated percentage of muscle mass using bioimpedance

OTHER OUTCOMES:
Weight | 8 weeks
  Body weight measured by kilograms
Waist circumference | 8 weeks
  Waist circumference measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Luis B Enríquez Sánchez, M.D., Study Director — Universidad Autonoma de Chihuahua
Locations (1):
- Hospital Central del Estado de Chihuahua, Chihuahua City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from this research study will be available if requested once the study is finalized.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available for up to five years since completion of the study.
Access Criteria: The request for the data will be by e-mail.